CLINICAL TRIAL: NCT03328468
Title: Development of Upper Limb Motor Scale "Awareness of Functional Tasks With Arm and Hand in Stroke"
Brief Title: Development of Upper Limb Motor Scale to Measure Quality of Movement and Body Awareness in Stroke
Acronym: AFAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PMR-2017-25877
Record Dates: First submitted 2017-10-19; First posted 2017-11-01 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Stroke
Keywords: Stroke
MeSH Terms: conditions — Stroke | interventions — Breathing Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breathing Exercise (Experimental)
  Interventions: Other: Breathing Exercise

INTERVENTIONS:
Other: Breathing Exercise — Breathing exercise for stroke patients

SUMMARY:
For the breathing intervention, participants completed two experimental sessions at least two weeks apart. The experimental sessions were randomized between the slow-breathing condition (6 breaths/min) or the control breathing condition (12 breaths/min). Breathing interventions were 15 minutes in length and completed with the assistance of the breathing app, Breathe Deep (Mineev, Bizi Apps LLC).

The breathing intervention is currently completed.

The reliability and validity study of AFAS is ongoing. This is a one-time visit for participants in which participants will undergo screening of sensation and movement as well as fill in some questionnaires.

DETAILED DESCRIPTION:
All participants had two visits for the breathing exercise. The only planned intervention was the breathing exercise, which is now concluded.

The protocol for the breathing intervention was as follows: The breathing protocol lasted 15 minutes. It was a guided breathing awareness session with a registered nurse (PhD student) who is also trained in integrative therapies and yoga instruction.

In parallel, during one of the visits the reliability and validity of a new scale for stroke to measure quality of movement and body awareness is tested.

This part is still ongoing and thus this becomes a one-time visit.

ELIGIBILITY:
Inclusion Criteria:

* Females and males ages 18-99 years of age
* People with stroke who are medically stable with one or more ischemic or
* hemorrhagic stroke(s)
* left or right hemiplegia
* willing and able to attend a one-time behavioral testing session
* willing and able to sign consent to participate
* able to hear, read and comprehend instructions given during the study
* English speaking (or willing to work with a (student) translator)

Exclusion Criteria:

* cognitive impairment (Mini-mental State Exam-brief version, <13/16)
* contractures in the tested arm that would hinder testing arm movements
* adults lacking capacity to consent
* severe neglect, aphasia, apraxia
* other medical conditions that preclude participation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2017-12-30 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Reliability of a new scale for stroke: Awareness of Functional Tasks with Arm and Hand in Stroke (AFAS scale) | Baseline
  AFAS contains 13 items
Validity a new motor scale for upper extremity Upper Limb Motor Scale in people with stroke (AFAS scale | Baseline
  Scale using 0-45 for measurement, 0 being low and 45 being high.

SECONDARY OUTCOMES:
Motor Evaluation Scale for Upper Extremity in Stroke Patients (MESUPES) | Baseline
  Scale using 0-58 for measurement, 0 being low and 58 being high. Assesses qualities of the arm and hand.
Revised Body Awareness Rating Scale (REVBA) | Baseline
  The Revised Body Awareness Rating Scales contains 12 items rated on a 4-point scale. Total scores range from 0 to 36 with lower scores indicating better body awareness.
Physical Body Experience Questionnaire (PBE) | Baseline
  The Physical Body Experience Questionnaire contains 12 items, rated on a 7-point Likert scale. Total scores range from 0 to 48 with lower scores indicated better physical body experience.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Van de Winckel, PhD, MS, PT, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.med.umn.edu/rehabmedicine/research/motor-scale-awareness